CLINICAL TRIAL: NCT07062029
Title: Can Laughter Heal the Spirit? The Impact of Laughter Yoga on Spiritual Well-Being and Spiritual Care Perception in Nursing Students
Brief Title: The Effect of Laughter Yoga on Spiritual Care Perception and Spiritual Well Being in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Begüm Güler, Research Assistant, Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/6-20
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Spirituality; Spiritual Well-being; Laughter Yoga
Keywords: Nursing; Spiritual- Well Being; spiritual care; laugther yoga
MeSH Terms: interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: This study was a randomized controlled trial with intervention and control groups. Sixty 3rd- and 4th-year nursing students provided informed consent and were randomized using randomizer.org and the URN method by drawing colored balls (green=intervention, white=control). The intervention group attended laughter yoga sessions twice a week for 4 weeks (each ~30 mins) led by a certified laughter yoga leader in a quiet, temperature-controlled lab suitable for movement. Sessions included warm-up, breathing, playful activities, and laughter exercises. Before the first session, students received an educational presentation and brochure. The control group received no intervention. Data were collected using the Spirituality and Spiritual Care Rating Scale and Three-Factor Spiritual Well-Being Scale 1 week before and 1 week after intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter Yoga Intervention (Experimental): Participants in this arm will attend laughter yoga sessions once a week for 4 weeks. Each session will last approximately 30 minutes and will be conducted by a certified laughter yoga leader in a quiet classroom environment where participants can move freely. The intervention aims to improve spiritual well-being and perception of spiritual care among nursing students.
  Interventions: Other: Laughter Yoga
- Control Group (No Intervention): Participants in this arm will not receive any intervention during the 4-week study period. They will complete the same pretest and posttest questionnaires as the intervention group, at the same time points, to evaluate their spiritual well-being and perception of spiritual care.

INTERVENTIONS:
Other: Laughter Yoga — The laughter yoga intervention consists of four sessions conducted once a week for four weeks. Each session lasts approximately 30 minutes and includes four components:
  * Warm-up exercises with clapping and rhythmic movements
  * Deep breathing exercises
  * Childlike playful activities and laughter exercises
  * Laughter meditation and relaxation Sessions are led by a certified laughter yoga leader in a quiet classroom setting that allows participants to move freely and comfortably. The intervention is designed to improve spiritual well-being and perception of spiritual care among nursing students.
  Arms: Laughter Yoga Intervention

SUMMARY:
The goal of this clinical trial is to learn if laughter yoga sessions improve spiritual well-being and perception of spiritual care among nursing students. The main questions it aims to answer are:

Does laughter yoga increase the spiritual well-being scores of participants? Does laughter yoga improve participants' perception of spiritual care? Researchers will compare laughter yoga to no intervention (control group) to see if laughter yoga has an effect on spiritual well-being and spiritual care perception.

Participants will:

Attend laughter yoga sessions once a week for 4 weeks (intervention group) Complete questionnaires about their spiritual well-being and perception of spiritual care before and after the intervention Control group will not receive any intervention during this period, but will complete the same questionnaires at the same time points

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the effects of laughter yoga on spiritual well-being and perception of spiritual care among nursing students. The study uses a pretest-posttest control group design. A total of 60 nursing students in their third and fourth years were randomly assigned to either the intervention group or the control group, with 30 students in each group.

The intervention group will participate in laughter yoga sessions once a week for 4 weeks. Each session will last approximately 30 minutes and will be conducted by a certified laughter yoga leader in a quiet classroom environment where students can move freely. The control group will not receive any intervention during the study period.

Spiritual well-being will be measured using the Spiritual Well-Being Scale (SWBS) and perception of spiritual care will be measured using the Spiritual Care-Giving Scale (SCGS). Both scales will be administered before the intervention (pretest) and after the 4-week intervention period (posttest).

The study hypothesizes that laughter yoga will significantly increase spiritual well-being scores and improve students' perception of spiritual care compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being a third- or fourth-year nursing student enrolled in the Faculty of Health Sciences, Department of Nursing at Izmir Demokrasi University during the 2024-2025 academic year
* Volunteering to participate in the study

Exclusion Criteria:

* Irregular attendance to the intervention sessions
* Failure to complete all sessions
* Voluntary withdrawal from the study
* Having a diagnosis of a respiratory disease (e.g., asthma, bronchitis, dyspnea)
* Having a diagnosis of inguinal hernia or epilepsy
* Having undergone abdominal surgery within the last three to six months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Change in Spiritual Well-Being Score | 1 week before intervention (baseline) and 1 week after completing the fourth session (Week 5)
  Spiritual well-being will be measured using the Three-Factor Spiritual Well-Being Scale, which has a total score range from 29 to 145, with higher scores indicating greater spiritual well-being.

SECONDARY OUTCOMES:
Change in Spirituality and Spiritual Care Rating Scale Score | 1 week before intervention (baseline) and 1 week after completing the fourth session (Week 5)
  Perception of spirituality and spiritual care will be assessed using the Spirituality and Spiritual Care Rating Scale, which is scored on a 1 to 5 scale, with higher scores indicating a more positive perception of spirituality and spiritual care.

CONTACTS AND LOCATIONS:
Overall Officials: Sadiye Associate Professor, PhD, Study Director — Izmir Democracy University
Locations (1):
- Izmir Democracy University, Izmir, Konak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the data are part of a thesis study with limited scope and there is no current plan or institutional repository available for data sharing. Additionally, participant privacy and confidentiality cannot be ensured for sharing de-identified data at this time.